CLINICAL TRIAL: NCT01403116
Title: Phase 3, Active-Controlled, Safety and Efficacy Trial of Oral Testosterone Undecanoate (TU) in Hypogonadal Men
Brief Title: Safety and Efficacy Trial of Oral Testosterone Undecanoate (TU) in Hypogonadal Men
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Clarus Therapeutics, Inc. (Industry)
Collaborators: PharmaNet (Industry); Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLAR-09007
Record Dates: First submitted 2011-07-25; First posted 2011-07-27 (Estimated); Results first posted 2018-08-14 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-07

CONDITIONS: Male Hypogonadism
Keywords: testosterone; male hypogonadism; low testosterone
MeSH Terms: conditions — Eunuchism | interventions — testosterone undecanoate; Coal Tar

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral testosterone undecanoate (TU) (Experimental): Treatment Period 1: 100 mg capsules, BID, with food
  Treatment Period 2: One of the following dosages:
  * 100 mg BID
  * 150 mg BID
  * 100 mg BID
  * 100 mg and 150 mg BID
  * 150 mg capsules BID
  Safety Follow-up Phase:
  Initial dose: ~84 doses Maintenance dose-Titrated dose: ~96 doses Safety follow-up at maintenance dose: ~540 doses
  Interventions: Drug: Oral testosterone undecanoate
- topical testosterone gel (Active Comparator): Treatment Period 1: 5 g of 1% transdermal T-gel applied QD
  Treatment Period 2:
  * 2.5 g of 1% transdermal T-gel applied QD
  * 5 g of 1% transdermal T-gel applied QD
  * 7.5 g of 1% transdermal T-gel applied QD
  * 10 g of 1% transdermal T-gel applied QD
  Safety Follow-up Phase:
  Initial dose: ~42 doses Maintenance dose-Titrated dose: ~48 doses Safety follow-up at maintenance dose: ~270 doses
  Interventions: Drug: topical testosterone gel

INTERVENTIONS:
Drug: Oral testosterone undecanoate — Starting dose: 200 mg T (as TU) BID. Doses may be titrated up to a maximum dose of 300 mg T (as TU) BID or down to a minimum dose of 100 mg T (as TU) BID based on serum T values collected at 4-6 hours post AM dose on Days 30 and 60.
  Other Names: Oral TU
  Arms: Oral testosterone undecanoate (TU)
Drug: topical testosterone gel — Starting dose: 5 g T applied once daily. Doses may be titrated up to a maximum dose of 10 g daily or down to a minimum dose of 2.5 g daily based on serum T values collected at 4-6 hours post AM dose on Days 30 and 60.
  Other Names: T-gel
  Arms: topical testosterone gel

SUMMARY:
The purpose of this study is to determine the safety and efficacy of an oral testosterone undecanoate formulation for use as testosterone-replacement therapy in men with low testosterone.

DETAILED DESCRIPTION:
This was a randomized, open-label, 2-arm, active controlled, 12-month study of Oral TU that planned to enroll ≈ 300 hypogonadal men (≈ 150/group) at multiple study sites. Incorporated in the design was dose titration based on serum T concentration assessed 4-6 hrs post AM dose. Following a 2-visit screening period during which a serum T concentration was measured, eligible subjects were randomized to either Oral TU (Group A) or transdermal T-gel (Group B) for dosing during Treatment Period 1 (Days 0 to 42). Group A was initially dosed with 400 mg T daily (two 100 mg capsules, orally, twice a day [BID]), and Group B was initially dosed with 5 g of transdermal 1% T-gel.

Serum T sampling was done on Day 30, 4-6 hours after the morning dose and these T concentration results were used to determine the need for dose titration. Dose titration occurred on Day 42 for Treatment Period 2, until Day 90. Subjects whose dose was titrated on Day 42 were re-evaluated on Day 60 , with dose adjustments made as necessary on Day 74.

Serum T sampling was performed on Day 90, for Oral TU subjects who had dose titration on Day 74, on Day 105. If the serum T level was > 1800 ng/dL, the sample was repeated; subjects were discontinued if the second assayed T concentration was > 1800 ng/dL. An additional dose titration was done for subjects whose Day 180 occurred after a protocol amendment. Subjects taking 150 mg T BID with serum T over 1500 ng/dL on two separate draws were discontinued.

Safety measures included physical examination, vital signs, fasting laboratory analysis (hematology, chemistry, urinalysis), CV biomarker monitoring [hs-CRP, Lp-PLA2, Lp(a), and ApoA1], measurement of sex hormone binding globulin (SHBG); luteinizing hormone (LH), follicle-stimulating hormone (FSH); prostate specific antigen (PSA), and the American Urological Association/International Prostate Symptom Score (AUA/I-PSS).

ELIGIBILITY:
Inclusion Criteria:

* Serum testosterone of less than or equal to 300 ng/dL on two occasions within one week (may wash out from previous oral, topical or buccal testosterone therapy)

Exclusion Criteria:

* Significant intercurrent disease of any type, in particular liver, kidney, uncontrolled or poorly controlled heart disease, or psychiatric illness
* Recent history of stroke, not including transient ischemic attack
* Untreated, sever obstructive sleep apnea.
* Hematocrit <35% or >48
* Serum transaminases >2 times upper limit of normal, serum bilirubin > 2.0 mg/dL and serum creatinine > 2.0 mgk/dL
* BMI > or equal to 36
* Stable doses of lipid-lowering medication for less than 3 months
* Stable doses of oral medication for diabetes for less than 2 months
* Abnormal prostate DRE [palpable nodule(s)], elevated PSA (>4 ng/mL), IPSS score > or equal to 19 points.
* History of breast cancer
* Use of dietary supplement saw palmetto or phytoestrogens and use of any dietary supplements that may increase serum testosterone within previous 4 weeks
* Known malabsorption syndrome and/or current treatment with oral lipase inhibitors
* History of abuse of alcohol or any drug substance within the previous 2 years
* Current use of antiandrogens, estrogens, oral CYP3A4 inducers or inhibitors, or long-acting opioid analgesics
* Receipt of any drug as part of a research study within 30 days of initial dose administration in this study.
* Blood donation within the 12 week period before the initial study dose.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2011-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Swerdloff, MD, Principal Investigator — Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Locations (30):
- United States (25):
  - Alabama Clinical Therapeutics, Inc., Birmingham, Alabama
  - Alabama Internal Medicine, PC, Birmingham, Alabama
  - Alabama Clinical Therapeutics, Calera, Alabama
  - Medical Affliated Research Center, Inc., Huntsville, Alabama
  - Quality of Life Medical and Research Centers, LLC, Tucson, Arizona
  - Providence Clinical Research, Burbank, California
  - South Orange County Endocrinology, Laguna Hills, California
  - Tower Urology, Los Angeles, California
  - David Geffen School of Medicine, Los Angeles, California
  - Harbor-UCLA Medical Center, LA Biomedical Research Institute, Torrance, California
  - Connecticut Clinical Research Center/ConnecTrials, Middlebury, Connecticut
  - University of CT School of Medicine, New Haven, Connecticut
  - South Florida Medical Research, Aventura, Florida
  - University of Louisville, Louisville, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - Boston University School of Medicine, Boston, Massachusetts
  - Maimonides Medical Center, Brooklyn, New York
  - Bruce R. Gilbert, MD, PhD, Great Neck, New York
  - University Urology Associates, New York, New York
  - Michael A. Werner, MD, PC, Purchase, New York
  - Sunstone Medical Research, Medford, Oregon
  - Urologic Consultants of Southeast Pennsylvania, Bala-Cynwyd, Pennsylvania
  - Research Across America, Carrollton, Texas
  - Research Across America, Dallas, Texas
  - University of Washington, Seattle, Washington
- Germany (5):
  - University of Bonn, Clinic for Dermatology and Allergy, Bonn
  - University of Halle, Center for Reproduction and Androlgoy, Halle
  - Praxis Dr. Szymula, Leipzig
  - Praxis Dr. Schulze, Markkleeberg
  - University of Muenster, Center for Reproduction and Andrology, Münster

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD

REFERENCES:
- [Derived] Honig S, Gittelman M, Kaminetsky J, Wang C, Amory JK, Rohowsky N, Dudley RE, Woun Seo B, Newmark J, Swerdloff R. Two-Year Analysis of a New Oral Testosterone Undecanoate (TU) Formulation in Hypogonadal Men: Efficacy, Impact on Psychosexual Function, and Safety. J Sex Med. 2022 Dec;19(12):1750-1758. doi: 10.1016/j.jsxm.2022.09.002. Epub 2022 Oct 20. PMID 36272969

RESULTS

PARTICIPANT FLOW:
Groups:
- Oral Testosterone Undecanoate (TU): Treatment Period 1: 100 mg capsules, BID, with food
  Treatment Period 2: One of the following dosages:
  * 100 mg BID
  * 150 mg BID
  * 100 mg BID
  * 100 mg and 150 mg BID
  * 150 mg capsules BID
  Safety Follow-up Phase:
  Initial dose: ~84 doses Maintenance dose-Titrated dose: ~96 doses Safety follow-up at maintenance dose: ~540 doses
  Oral testosterone undecanoate: Starting dose: 200 mg T (as TU) BID. Doses may be titrated up to a maximum dose of 300 mg T (as TU) BID or down to a minimum dose of 100 mg T (as TU) BID based on serum T values collected at 4-6 hours post AM dose on Days 30 and 60.
- Topical Testosterone Gel: Treatment Period 1: 5 g of 1% transdermal T-gel applied QD
  Treatment Period 2:
  * 2.5 g of 1% transdermal T-gel applied QD
  * 5 g of 1% transdermal T-gel applied QD
  * 7.5 g of 1% transdermal T-gel applied QD
  * 10 g of 1% transdermal T-gel applied QD
  Safety Follow-up Phase:
  Initial dose: ~42 doses Maintenance dose-Titrated dose: ~48 doses Safety follow-up at maintenance dose: ~270 doses
  topical testosterone gel: Starting dose: 5 g T applied once daily. Doses may be titrated up to a maximum dose of 10 g daily or down to a minimum dose of 2.5 g daily based on serum T values collected at 4-6 hours post AM dose on Days 30 and 60.
Period: Overall Study
Arm/Group | Oral Testosterone Undecanoate (TU) | Topical Testosterone Gel
Started | 161 | 160
Randomized | 162 | 163
Randomized in Error/ No Treatment Recvd | 1 | 3
Completed | 129 | 133
Not Completed | 32 | 27
Not completed — Adverse Event | 7 | 4
Not completed — Lost to Follow-up | 7 | 5
Not completed — Withdrawal by Subject | 12 | 15
Not completed — Non-compliance of study drug | 3 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — undisclosed Hx of Prostate Ca | 1 | 0
Not completed — Hct >54% | 2 | 0
Not completed — unable to keep appointments | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Testosterone Undecanoate (TU) | Topical Testosterone Gel | Total
Number analyzed (Participants) | 161 | 160 | 321
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 134 | 136 | 270
  >=65 years | 27 | 24 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (11.06) | 54.7 (11.18) | 54.9 (11.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 161 | 160 | 321
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 141 | 143 | 284
  Germany | 20 | 17 | 37

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Treated Patients With Average Serum Testosterone (T) Concentrations (Cavg) Between 300 and 1000 ng/dL
Description: The percentages of treated subjects that had 24-hour serum testosterone (T) average concentrations (Cavg) between 300 and 1000 ng/dL
Time Frame: Following 90 days of treatment
Population: Intent to treat population
Measure: Geometric Mean (95% Confidence Interval); unit: percentage of partipants
Arm/Group | Oral Testosterone Undecanoate (TU) | Topical Testosterone Gel
Number analyzed (Participants) | 146 | 149
percentage of partipants | 83.6 [76.5 to 89.2] | 79.2 [71.8 to 85.4]

2. Secondary Outcome: % of Oral TU Subjects With 24-hour Maximum Serum T Concentrations (Cmax) Greater Than 1500 ng/dL on Day 90
Description: Percentage of Oral TU treated patients who reached study day 90 and had a maximum serum T concentrations (Cmax) values greater than 1500 ng/dL(objective to meet <15%).
Time Frame: 90 days
Population: Percent of oral TU treated subjects with Cmax >1500 ng/dL at Study Day 90
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Testosterone Undecanoate (TU)
Number analyzed (Participants) | 149
Participants | 61

ADVERSE EVENTS:
Arm/Group | Oral Testosterone Undecanoate (TU) | Topical Testosterone Gel
All-Cause Mortality (participants affected / at risk) | 0/161 | 0/160
Serious Adverse Events (participants affected / at risk) | 11/161 | 6/160
Other Adverse Events (participants affected / at risk) | 110/161 | 82/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Testosterone Undecanoate (TU) (N=161) | Topical Testosterone Gel (N=160)
Acute myocardial infarction (Cardiac disorders) | 2 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Coronary Artery Disease (Cardiac disorders) | 2 | 1
Appendicitis (Infections and infestations) | 0 | 2
Gastroenteritis (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Brachial plexus injury (Injury, poisoning and procedural complications) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Inverterbral disc degeneration (Musculoskeletal and connective tissue disorders) | 3 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 0
Nervous system disorder (Nervous system disorders) | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Testosterone Undecanoate (TU) (N=161) | Topical Testosterone Gel (N=160)
Polycythaemia (Blood and lymphatic system disorders) | 13 | 6
Abdominal discomfort (Gastrointestinal disorders) | 5 | 0
Diarrhea (Gastrointestinal disorders) | 9 | 3
Eructation (Gastrointestinal disorders) | 4 | 0
Nausea (Gastrointestinal disorders) | 4 | 4
Oedema peripheral (General disorders) | 9 | 2
Gastroenteritis viral (Infections and infestations) | 4 | 2
Nasopharyngitis (Infections and infestations) | 10 | 7
Sinusitis (Infections and infestations) | 5 | 5
Upper respiratory tract infection (Infections and infestations) | 11 | 4
Prostatic specific antigen (Investigations) | 5 | 8
Arthalgia (Musculoskeletal and connective tissue disorders) | 4 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Dizziness (Nervous system disorders) | 4 | 2
Headache (Nervous system disorders) | 4 | 5
Prostatitis (Reproductive system and breast disorders) | 4 | 2
Prostatomegaly (Reproductive system and breast disorders) | 9 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Acne (Skin and subcutaneous tissue disorders) | 1 | 4
Hypertension (Vascular disorders) | 6 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days